CLINICAL TRIAL: NCT02416778
Title: Effect of Intravenous Iron (Ferinject®) on Exercise Capacity and Quality of Life of Stable COPD Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georg-Christian Funk (Other)
Responsible Party: Sponsor-Investigator, Georg-Christian Funk, M.D., Assoc. Prof., Otto Wagner Hospital
Organization: Otto Wagner Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Iron-COPD Pilotstudy
Record Dates: First submitted 2015-02-10; First posted 2015-04-15 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Iron deficiency; 6 Minute-Walking-Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Iron Deficiencies | interventions — ferric carboxymaltose; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Ferric carboxymaltose, Ferinject® 50mg Iron/ml Solution for Injection / Infusion will be administered in patients with COPD
  Interventions: Drug: Ferric carboxymaltose, Ferinject® 50mg Iron/ml Solution for Injection / Infusion

INTERVENTIONS:
Drug: Ferric carboxymaltose, Ferinject® 50mg Iron/ml Solution for Injection / Infusion

SUMMARY:
Disordered iron metabolism characterizes an important determinant of impaired exercise tolerance and work capacity. Iron-deficiency anemia commonly features impaired aerobic capacity caused by decreased oxygen carrying capacity, and has been associated with a negative effect on dyspnea and walking distance.

Apart from that, iron deficiency without anemia was shown to affect endurance and energetic efficiency via decreased tissue oxidative capacity. Consequently, depleted iron stores could be capable of causing fatigue, breathlessness and impaired exercise tolerance, which are common features of chronic cardiopulmonary diseases like chronic heart failure (CHF) and COPD (Chronic Obstructive Pulmonary Disease). Indeed, a current surge of interest aimed at potential underlying determinants in CHF and COPD independent of the primarily disordered organ.

Recent studies identified iron deficiency without anemia as an independent factor of reduced exercise intolerance in CHF as well as in COPD. Moreover, intravenous iron application significantly improved exercise capacity in CHF patients with iron deficiency in presence as well as in absence of anemia. Comparable to CHF, the daily living of patients with COPD is compromised by impaired exercise tolerance.

However, airflow limitation, as the foremost characteristic of COPD shows only weak associations with exercise capacity. In line with that, exercise capacity showed no remarkable improvement in lung transplant recipients, underlining the presence of systemic determinants of limited exercise tolerance like iron deficiency. The investigators showed that iron deficiency is present in 50% of stable COPD patients (unpublished data), which is according to recently published data.

The investigators presume that iron deficiency contributes to limited exercise capacity in COPD patients. Thus, the aim of this study is to determine whether iv iron is associated with increases exercise capacity in COPD.

Therefore the investigators hypothesize that filling up depleted iron storages will increase exercise capacity, measured by the 6-MWT (Minute Walking Test).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease according to the current guidelines
* Evidence of irreversible airflow obstruction on spirometry (i.e. an increase of less than 200ml and 15% in the post-bronchodilator FEV1)
* 30% < FEV1 < 80% predicted
* Stable COPD medication: no dose changes in COPD medication within last 4 weeks
* Age of 40 to 75 years
* Body mass index < 30 kg/m2
* Iron deficiency:

ferritin <100 ng/mL or ferritin 100-300 ng/mL when TSAT (Transferrin saturation) <20%

* Hb between 9.5 and 13.5 g/dL
* MMRC (Modified Medical Research Council Scale) 0 to 3
* Patient must be able to perform the bicycle exercise test according to investigator

Exclusion Criteria:

* Meeting contraindications of iv iron administration
* Known active infection
* C-reactive protein>20 mg/L
* clinically significant bleeding
* active malignancy
* History of congestive heart failure
* BNP (Brain Natriuretic Peptide) ≥ 250 pg/ml
* Evidence of myocardial ischemia during Cardiopulmonary Exercise Test (CPET) (i.e. chest pain or signs of ischemia in ECG)
* uncontrolled Hypertension
* other clinical significant chronic heart disease
* Acute myocardial infarction or acute coronary syndrome, transient ischaemic attack or stroke within the last 3 months
* History of peripheral artery occlusive disease
* Typical claudication
* Anaemia due to reasons other than iron deficiency (e.g.haemoglobinopathy)
* History of erythropoietin, i.v. or oral iron therapy, and blood transfusion in previous 12 weeks and/or such therapy planned within the next 6 months
* Immunosuppressive therapy or renal dialysis
* ALT (Alanine Aminotransferase) or AST (Aspartate Aminotransferase) >3times upper limit of normal
* Hemochromatosis
* Significant lung diseases other than COPD
* pulmonary hypertension (maximum of velocity tricuspid regurgitation > 2,8m/sec)
* Exacerbation within prior 4 weeks
* > 1 exacerbation within last year
* bronchoscopic lung volume reduction (BLVR)
* Malignancy within the past 5 years
* Autoimmune diseases
* Rheumatoid diseases
* Chronic renal failure (defined through: eGFR (Estimated Glomerular Filtration Rate) < 60 ml/min)
* Active diet
* Physical rehabilitation training
* Pregnancy, breast feeding
* Participation in other therapeutic trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoint: Increased exercise capacity in 6-Minute-Walking-Test (walking distance in meters [m]) | Study week 12
Efficacy Endpoint: Cardiopulmonary Exercise Test (FEV1 [ml] / FVC [% predicted]) | Study week 12

SECONDARY OUTCOMES:
Tolerability/Safety Endpoint: Acute COPD exacerbation | Pre-Screening, Study Day 0, Study week1, study week 4, study week 8 and study week 12
Adverse events of iron administration | Pre-Screening, Study Day 0, Study week1, study week 4, study week 8 and study week 12

CONTACTS AND LOCATIONS:
Overall Officials: Georg-Christian Funk, M.D.Ass.Prof, Principal Investigator — Otto Wagner Spital, Dep. of Respiratory and Critical Care Medicine, Pavillon Hermann, Sanatoriumstr. 2, A-1140 Vienna
Locations (1):
- Otto Wagner Spital, Dep. of Respiratory and Critical Care Medicine, Vienna, Vienna, Austria